CLINICAL TRIAL: NCT04834258
Title: What Happens to Pulmonary Function and Functional Exercise Capacity When Walking Training is Combined With Respiratory Muscle Training in Patients With Parkinson's Disease: A Randomized Double-blind Controlled Trial
Brief Title: Effects of Walking and Respiratory Muscle Training on Pulmonary Function and Functional Exercise Capacity in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5562
Record Dates: First submitted 2021-03-28; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: walking training; respiratory muscle training; pulmonary function; functional capacity
MeSH Terms: conditions — Parkinson Disease | interventions — Walking; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Outcomes Assessor (PFT, PImax, PEmax, SNIP, 6MWT, UPDRS III): Blind to group allocation Investigator: Blind to initial and final assessments Participant: Blind to training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking and respiratory muscle training group (Experimental): Walking and respiratory muscle training group (W+ RMT) received walking training in addition to respiratory muscle training for a period of 8 weeks.
  Walking training was performed at least 5 days a week, twice a day, for 15 min. Walking distance was calculated according to patients' 6 minute walking distance.
  Respiratory muscle training was performed using the threshold loading method as inspiratory and expiratory muscle training. This training was applied at least 5 days per week, twice a day, 15 minutes each session. (15 minutes inspiratory muscle training + 15 minutes expiratory muscle training). A Threshold Inspiratory Muscle Trainer (IMT) and threshold positive expiratory pressure (Threshold PEP) were used for the training.
  Patients were called for the hospital once a week to asses mouth pressure and 6 minute walking test (6 MWT) and their training intensity was arranged.
  Interventions: Other: Walking and respiratory training
- Respiratory muscle training group (Active Comparator): In the Respiratory muscle training group (RMT), Respiratory muscle training was performed using the threshold loading method as inspiratory and expiratory muscle training. This training was applied at least 5 days per week, twice a day, 15 minutes each session. (15 minutes inspiratory muscle training + 15 minutes expiratory muscle training). A Threshold Inspiratory Muscle Trainer (IMT) and threshold positive expiratory pressure (Threshold PEP) were used for the training. Patients were called for the hospital once a week to asses mouth pressure and their training intensity was arranged
  Interventions: Other: Respiratory muscle training

INTERVENTIONS:
Other: Walking and respiratory training — Walking and respiratory muscle training group ( W+ RMT) received walking training in addition to respiratory muscle training for a period of 8 weeks.
  Walking training was performed at least 5 days a week, twice a day, for 15 min. Walking distance was calculated according to patients' 6 minute walking distance.
  Respiratory muscle training was performed using the threshold loading method as inspiratory and expiratory muscle training. This training was applied at least 5 days per week, twice a day, 15 minutes each session. (15 minutes inspiratory muscle training + 15 minutes expiratory muscle training). A Threshold Inspiratory Muscle Trainer (IMT) and threshold positive expiratory pressure (Threshold PEP) were used for the training.
  Patients were called for the hospital once a week to asses mouth pressure and 6 minute walking test (6 MWT) and their training intensity was arranged
  Other Names: Respiratory muscle training device and exercise program
  Arms: Walking and respiratory muscle training group
Other: Respiratory muscle training — In the Respiratory muscle training group, Respiratory muscle training was performed using the threshold loading method as inspiratory and expiratory muscle training. This training was applied at least 5 days per week, twice a day, 15 minutes each session. (15 minutes inspiratory muscle training + 15 minutes expiratory muscle training). A Threshold Inspiratory Muscle Trainer (IMT) and threshold positive expiratory pressure (Threshold PEP) were used for the training. Patients were called for the hospital once a week to asses mouth pressure and their training intensity was arranged.
  Other Names: Respiratory muscle training device
  Arms: Respiratory muscle training group

SUMMARY:
The purpose of this randomised and controlled study is to investigate the effects of walking training combined with respiratory muscle training on pulmonary function, respiratory muscle strength, and functional exercise capacity.

DETAILED DESCRIPTION:
Although respiratory dysfunction has been recognized as a cause of morbidity and mortality in patients with Parkinson's disease (PD), most of the patients were not aware of their respiratory problems due to restriction in their activities.

Respiratory dysfunction in patients with PD has not been well characterized. However, there are many studies showing restrictive or obstructive type respiratory disorders and decreased respiratory muscle strength in the literature. Ineffective cough due to decreased respiratory muscle strength may cause to secretion retention and secondary infections in PD patients who have severe symptoms. Therefore, the assessment and rehabilitation of these respiratory problems is important in PD patients treatment. There are studies in the literature showing that respiratory muscle training is effective in PD.

Walking difficulty is seen as a common problem in PD. Typically, walking is slow despite adequate Levodopa therapy. It is known that exercise capacity may be affected by respiratory impairment, walking difficulties and personal exercise habits in patients with PD. Respiratory and walking problems lead to limitation of physical activity in PD, which leads to a decrease in exercise capacity. In a recently published article reported that walking is a good example of exercise.

Although walking training is important for PD patients, there is no studies what happens to pulmonary function and functional exercise capacity when walking training is combined with respiratory muscle training in patients with Parkinson's disease. Therefore, this study planned to investigate the effects of walking and respiratory muscle training on pulmonary function and functional exercise capacity in PD.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed according with PD to the clinical criteria of the United Kingdom Parkinson's Disease Society Brain Bank diagnostic criteria
* being in phase 1-3 according to the Hoehn-Yahr (H-Y) scale,
* being under anti-parkinson's treatment, and
* being in the "on"period.

Exclusion Criteria:

* • dyskinesia, (which may be obstacles to the tests),

  * chronic respiratory disease,
  * dementia,
  * co-operation difficulty,
  * cognitive impairment (mini-mental test score <24), and
  * other neurologic, cardiovascular or musculoskeletal problems that impede walking.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2011-08-10 (Actual); Study Completion 2011-09-15 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory mouth pressure (PImax) and Maximal Expiratory mouth pressure (PEmax) | Change from baseline maximal inspiratory mouth pressure and maximal expiratory pressure at 8 weeks
  Maximum inspiratory pressure (PImax) is the classic volitional test for inspiratory muscle strength. It is measured as the highest mouth pressure (cmH2O) sustained for 1 s during a maximum inspiratory effort against a quasi occlusion. Assessment is carried out according to the Black and Hyatt technique.
  Maximum expiratory pressure (PEmax) is the classic volitional test for expiratory muscle strength. It is measured as the highest mouth pressure (cmH2O) sustained for 1 s during a maximum expiratory effort against a quasi occlusion. Assessment is carried out according to the Black and Hyatt technique.
Functional Exercise Capacity | Change from baseline functional exercise capacity at week 8
  Functional exercise capacity was measured with the 6 Minute Walk Test (6MWT) according to the American Thoracic Society (ATS) guidelines. The 6 minutes walking distance (6MWD) was recorded in meters.

SECONDARY OUTCOMES:
Spirometric measurements | Baseline and week 8
  Forced expiratory volume in one second (FEV1),Forced Vital Capacity (FVC),FEV1/FVC ratio were measured.
Unified Parkinson's Disease Rating Scale - motor examination | Baseline and week 8
  Unified Parkinson's Disease Rating Scale - motor examination (UPDRS- III) of the scale assesses the motor signs of Parkinson's disease.All items must have an integer rating (no half points, no missing ratings). Specific instructions are provided for the testing of each item. The motor UPDRS consists of five-category ordinal items scored 0-4.The total motor UPDRS exam score ranges from 0 to 108. A higher scores indicating greater disability.

OTHER OUTCOMES:
Sniff nasal inspiratory pressure (SNIP) | Baseline and week 8
  Sniff nasal inspiratory pressure (SNIP) measurement is a volitional noninvasive assessment of inspiratory muscle strength. A maximum of 10 sniffs is generally used. It is a simple procedure consisting of measuring peak nasal pressure (cmH2O) as a result of maximal sniff performance through from the end of expiration with the open nostril while the the other one is closed.

CONTACTS AND LOCATIONS:
Overall Officials: Semra OGUZ, PhD, Principal Investigator — Marmara University; Nilgun Gurses, Prof., Study Director — Bezmialem Vakif University; Hulya Apaydin, Prof, Study Chair — Istanbul University - Cerrahpasa

REFERENCES:
- [Background] Baille G, De Jesus AM, Perez T, Devos D, Dujardin K, Charley CM, Defebvre L, Moreau C. Ventilatory Dysfunction in Parkinson's Disease. J Parkinsons Dis. 2016 Jun 16;6(3):463-71. doi: 10.3233/JPD-160804. PMID 27314755
- [Background] Sabate M, Rodriguez M, Mendez E, Enriquez E, Gonzalez I. Obstructive and restrictive pulmonary dysfunction increases disability in Parkinson disease. Arch Phys Med Rehabil. 1996 Jan;77(1):29-34. doi: 10.1016/s0003-9993(96)90216-6. PMID 8554470
- [Background] Canning CG, Alison JA, Allen NE, Groeller H. Parkinson's disease: an investigation of exercise capacity, respiratory function, and gait. Arch Phys Med Rehabil. 1997 Feb;78(2):199-207. doi: 10.1016/s0003-9993(97)90264-1. PMID 9041903
- [Background] Saleem AF, Sapienza CM, Okun MS. Respiratory muscle strength training: treatment and response duration in a patient with early idiopathic Parkinson's disease. NeuroRehabilitation. 2005;20(4):323-33. PMID 16403998
- [Background] Rodriguez MA, Crespo I, Del Valle M, Olmedillas H. Should respiratory muscle training be part of the treatment of Parkinson's disease? A systematic review of randomized controlled trials. Clin Rehabil. 2020 Apr;34(4):429-437. doi: 10.1177/0269215519896054. Epub 2019 Dec 26. PMID 31875689
- [Background] Alves WM, Alves TG, Ferreira RM, Lima TA, Pimentel CP, Sousa EC, Abrahin O, Alves EA. Strength training improves the respiratory muscle strength and quality of life of elderly with Parkinson disease. J Sports Med Phys Fitness. 2019 Oct;59(10):1756-1762. doi: 10.23736/S0022-4707.19.09509-4. Epub 2019 May 20. PMID 31113177
- [Background] Koseoglu F, Inan L, Ozel S, Deviren SD, Karabiyikoglu G, Yorgancioglu R, Atasoy T, Ozturk A. The effects of a pulmonary rehabilitation program on pulmonary function tests and exercise tolerance in patients with Parkinson's disease. Funct Neurol. 1997 Nov-Dec;12(6):319-25. PMID 9503194